CLINICAL TRIAL: NCT01929577
Title: A Phase 1, Single-Dose, Open-Label, 3-Period, Randomized Crossover Study to Assess the Relative Bioavailability Between Two ASP015K Tablet Formulations and the Food Effect on a New Tablet Formulation in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability Between Two ASP015K Tablets and the Food Effect of a New Tablet in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 015K-CL-PK09
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Bioavailability of ASP015K; Healthy Subjects; Pharmacokinetics of ASP015K; Food Effect of ASP015K
Keywords: ASP015K; healthy subjects
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP015K Test Tablet - Fasting Conditions (Experimental): ASP015K administered as a single tablet under fasting conditions.
  Interventions: Drug: ASP015K
- ASP015K Reference Tablet - Fasting Conditions (Experimental): ASP015K administered via multiple tablets under fasting conditions
  Interventions: Drug: ASP015K
- ASP015K Test Tablet -Fed Conditions (Experimental): ASP015K administered as a single tablet under fed conditions
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — oral tablet

SUMMARY:
The purpose of this study is to determine the relative bioavailability of ASP015K under fasting conditions after single-dose administration between a test-tablet formulation and a reference-tablet formulation. This study will also evaluate the food effect on bioavailability of the test formulation, and evaluate the safety and tolerability after single-dose administration of the test- and reference-tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must be of non-childbearing potential (i.e., post-menopausal [defined as at least 1 year without menses prior to screening], or documented surgically sterile or status post hysterectomy [at least 1 month prior to screening]).
* Female subject must have a negative pregnancy test at screening and day -1 of treatment period 1.
* Female subject must not donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at screening and continue throughout the study period and for 90 days after final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after final study drug administration.
* Subject has a Body Mass Index (BMI) range of 18.5-32.0 kg/m2, inclusive, and must weigh at least 50 kg at screening.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months before screening assessment or breast feeding within 3 months before screening.
* Subject has a known or suspected hypersensitivity to ASP015K, or any components of the formulation used.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to first clinic check-in.
* Subject has used any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, with the exception of hormone replacement therapy (HRT), intermittent acetaminophen (to a maximum of 2 g/day).
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months prior to screening.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits) prior to day -1 of treatment period 1.
* Subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic check-in on day -1 of treatment period 1.
* Subject has a positive test for hepatitis B surface antigen (HBsAg), anti-hepatitis A virus (HAV) (Immunoglobulin [Ig] M), anti-hepatitis C virus (HCV), hepatitis B core antibody, or anti-human immunodeficiency virus (HIV) type 1 or type 2 at screening.
* Subject has a positive tuberculosis (TB) skin test, Quantiferon Gold® test or T-SPOT® test at screening.
* Subject received any vaccine within 60 days prior to study drug administration.
* Subject has an absolute neutrophil count (ANC) < 2000 cells/mm3 or a creatine phosphokinase (CPK) > 1.5 x ULN at screening or day -1 of treatment period 1.
* Subject has had major gastrointestinal (GI) surgery or has a medical condition, which may inhibit the absorption and/or metabolism of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASP015K: Cmax | Day 1-4 of each treatment period
  Maximum Concentration (Cmax)
Pharmacokinetic parameter of ASP015K: AUClast | Day 1-4 of each treatment period
  Area Under the Curve from time zero to the last measurable time (AUClast)
Pharmacokinetic parameter of ASP015K: AUCinf | Day 1-4 of each treatment period
  Area Under the Curve from time zero extrapolated to infinity (AUCinf)

SECONDARY OUTCOMES:
Composite of pharmacokinetic parameters of ASP015K: tmax, t1/2 | Day 1-4 of each treatment period
  Time to Maximum Concentration (tmax), apparent terminal elimination half-life (t1/2)
Composite of pharmacokinetic parameters of ASP015K metabolites: Cmax, AUClast, AUCinf, tmax, t1/2 | Day 1-4 of each treatment period
Safety assessed by adverse events, clinical laboratory evaluations, 12-lead ECG measurements, physical examinations and vital sign measurements | Up to Day 4 in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel - Early Phase Clinical Unit, Baltimore, Maryland, United States